CLINICAL TRIAL: NCT05753852
Title: Open Label Extension Study to Investigate Long Term Safety, Tolerability and Efficacy of Tauroursodeoxycholic Acid in Patients With ALS Who Completed the TUDCA-ALS Study
Brief Title: Open Label Extension of TUDCA-ALS Study
Acronym: TUDCA-ALS OLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Humanitas Mirasole SpA (Other)
Collaborators: University of Ulm (Other); University of Sheffield (Other); University Hospital, Tours (Other); KU Leuven (Other); UMC Utrecht (Other); University of Dublin, Trinity College (Other); Bruschettini S.r.l. (Unknown); Istituto Superiore di Sanità (Other); Motor Neurone Disease Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2020/755094/2017/OLE
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Bile acids; Deoxycholic Acid
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ursodoxicoltaurine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental)
  Interventions: Drug: Tauroursodeoxycholic Acid

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid — Tauroursodeoxycholic acid (TUDCA) 250 mg capsules Doses: 4 capsules (1 g) twice daily 10-15 minutes after a meal Mode of administration: orally Duration: 18 months
  Other Names: TUDCA,Tudcabil, Taurolite

SUMMARY:
This study will provide extended access to patients and assess longer-term outcomes on patients who have completed the TUDCA-ALS study.

DETAILED DESCRIPTION:
The TUDCA-ALS Open label extension study is designed to investigate long term safety, tolerability and efficacy of tauroursodeoxycholic acid in patients with ALS who completed the TUDCA-ALS study

ELIGIBILITY:
Inclusion Criteria:

* Completion of the visit M18 (Month 18) of the TUDCA-ALS clinical trial.
* Signed informed consent for participation in the TUDCA-ALS Extension sub-study

Exclusion Criteria:

* Treatment with edaravone or other unaccepted concomitant therapy
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive TUDCA or that the subject is unable or unlikely to comply with the dosing schedule or study evaluations
* The patient of reproductive potential is sexually active and is not willing to use highly effective contraception during the study and up to 90 days after the day of last dose
* The patient is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and tolerability of TUDCA during the open-label phase | 18 months
  Long-term safety and tolerability assessed through adverse reaction, concomitant treatment, and routine biochemistry analyses

SECONDARY OUTCOMES:
Survival time | 18 months
  Survival time measured by death or respiratory insufficiency (defined as tracheostomy or the use of non-invasive ventilation for ≥22 h per day for ≥10 consecutive days).
Change in disease progression and functional impairment | 18 months
  Change in disease progression and functional impairment as measured by ALSFRS-R.

CONTACTS AND LOCATIONS:
Locations (23):
- Katholieke Universiteit Leuven, Leuven, Belgium
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire Limoges, Limoges
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Regional Universitaire de Tours, Tours
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universität Ulm, Ulm
- Trinity College Dublin, Dublin, Ireland
- Italy (6):
  - IRCCS Istituto Auxologico Italiano, Milan
  - NEuroMuscular Omnicentre. Fondazione Serena Onlus, Milan
  - AOU Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - AOU Città della Salute e della Scienza di Torino, Torino
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- United Kingdom (5):
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Plymouth Hospitals NHS Trust, Plymouth
  - Salford Royal NHS Foundation Trust, Salford
  - University of Sheffield, Sheffield
  - Royal Stoke University Hospital, Stoke